CLINICAL TRIAL: NCT02461069
Title: A 24-week, Multicenter, Exploratory, Two Arm Study to Assess the Effect of Dimethyl Fumarate on Immune-Modulatory Action on T Cells in Patients With Relapsing Remitting Multiple Sclerosis (DIMAT-MS)
Brief Title: Investigation of the Effect of Dimethyl Fumarate on T Cells in Patients With Relapsing Remitting Multiple Sclerosis
Acronym: DIMAT-MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DIMAT-MS; 2014-003481-25 (EudraCT Number); U1111-1164-2476 (Other: Universal Trial Number)
Record Dates: First submitted 2015-05-27; First posted 2015-06-03 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: dimethyl fumarate
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dimethyl fumarate treatment arm (A) (Active Comparator): All patients will receive dimethyl fumarate (Tecfidera®) according to national recommendations (Krankheitsbezogenes Kompetenznetz Multiple Sklerose, KKNMS) from week 0 to week 24 (EOS-1) in the core study.
  Interventions: Drug: Dimethyl fumarate
- Healthy subject arm (B) (No Intervention): Healthy subjects will not receive any treatment for RRMS during the study.

INTERVENTIONS:
Drug: Dimethyl fumarate — Dimethyl fumarate (Tecfidera®) treatment is initiated by daily administration of 120 mg Tecfidera® p.o. in the morning in week 0. At week 1, the dose is increased to 120 mg Tecfidera® p.o. twice daily, split into a morning and an evening dose. At week 2, the daily dose is further increased to 240 mg Tecfidera® p.o. in the morning and 120 mg Tecfidera® p.o. in the evening. Finally at week 3, the dose will be increased to the final daily dose of 240 mg Tecfidera® p.o. in the morning and 240 mg Tecfidera® p.o. in the evening and maintained throughout the study.
  Other Names: Tecfidera®
  Arms: Dimethyl fumarate treatment arm (A)

SUMMARY:
This is an exploratory study, which allows analysis of multiple immune parameters derived from peripheral blood mononuclear cells (PBMCs) from patients with relapsing remitting multiple sclerosis before and during immune-modulatory treatment with dimethyl fumarate in comparison to PBMCs from healthy subjects.

DETAILED DESCRIPTION:
The purpose of the trial is to shed more light on the mechanisms of action of dimethyl fumarate in patients with relapsing remitting multiple sclerosis. More specifically the influence of dimethyl fumarate on peripheral immune cells will be addressed to evaluate changes in cytokine production by the distinct T cell subsets and the differentiation capacity of naïve T cells. Furthermore, the impact of dimethyl fumarate treatment on the migratory capacity of T cells as well as the evaluation of changes in the suppressive capacity of regulatory T cells will be evaluated. To put the obtained results into context, response data of dimethyl fumarate-treated patients will be compared with data from healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* H-1. Written informed consent must be obtained before any assessment is performed.
* H-2. Male and female subjects aged 18 - 60 years.
* H-3. No history of multiple sclerosis or clinically isolated syndrome.
* H-4. No history of other autoimmune diseases, which has been treated systemically with corticosteroids, immunomodulators or immunosuppressive drugs at any time point.

RRMS patients:

* MS-1. Written informed consent must be obtained before any assessment is performed.
* MS-2. Male and female subjects aged 18 - 60 years.
* MS-3. Patients with RRMS, defined by 2010 revised McDonald criteria.
* MS-4. Patients with an Expanded Disability Status Scale (EDSS) score of 0-6.0.
* MS-5. Patients with one of the following treatment status:

  * Naïve to disease modifying (DM) treatment (i.e. no DM treatment for at least 1 month),
  * Currently on MS therapy with interferon β-1 or glatiramer acetate and willing to switch to dimethyl fumarate (Tecfidera®).
* MS-6. MRI-scan of the brain ≤ 3 months at screening.

Exclusion Criteria:

RRMS patients:

* MS-1. Known hypersensitivity to dimethyl fumarate or any ingredients of Tecfidera® (microcrystalline cellulose; croscarmellose-sodium; talcum; high dispersion, hydrophobic silicon dioxide; magnesiumstearate (Ph. Eur.); triethylcitrate; methacrylic acid-methacrylate copolymer (1:1) (Ph. Eur.); methacrylic acid-ethylacrylate copolymer (1:1)-dispersion 30% (Ph. Eur.), simeticon, sodiumdodecylsulfate, polysorbate 80, gelantine, titanium oxide (E171), brilliant blue (E133), hydrated Iron(III)-oxide hydroxide (E172), shellac, potassium hydroxide.
* MS-2. A MS-relapse within 30 days prior to screening.
* MS-3. Known history of active tuberculosis or active tuberculosis determined by a positive QuantiFERON® TB Gold test (i.e. a negative test result has to be provided at screening unless a negative test result exists from the last 3 months prior to screening).
* MS-4. Moderate to severe impairment of liver function or persisting elevations > 2 x ULN (confirmed by retest) of serum glutamic pyruvic transaminase/ alanine aminotransferase (SGPT/ALT) or serum glutamic oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST), except patients with confirmed Gilbert´s syndrome (Meulengracht´s disease).
* MS-5. Moderate to severe impairment of renal function, as shown by serum creatinine > 133 μmol/L (or > 1.5 mg/dL).
* MS-6. Patients with significantly impaired bone marrow function or significant anemia, leukopenia, neutropenia or thrombocytopenia.
* MS-7. Women of childbearing potential not utilizing highly effective contraception.

Both populations:

* MS/H-1. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* MS/H-2. Subjects unlikely to comply with protocol as determined by investigator, e.g., uncooperative attitude, inability to return for follow-up visits (e.g. major physical disability), and known unlikelihood of completing the study.
* MS/H-3. Clinically relevant cardiovascular, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the subject at risk by participating in the study.
* MS/H-4. Subjects with ulcerative colitis or Crohn´s disease.
* MS/H-5. Subjects with a congenital or acquired severe immunodeficiency, a history of cancer (except for basal or squamous cell skin lesions which have been surgically excised, with no evidence of metastasis), lymph proliferative disease, or any subject who has received lymphoid irradiation.
* MS/H-6. Human immunodeficiency virus (HIV) positive, hepatitis B virus positive or hepatitis C virus positive subjects (i.e. a negative test result has to be provided at screening. In the presence of a negative test result from the last 3 months prior to screening, the test has not to be repeated at screening.).
* MS/H-7. Acute or chronic infection.
* MS/H-8. History of drug or alcohol abuse.
* MS/H-9. Use of adrenocorticotrophic hormone (ACTH) or systemic corticosteroids for 4 weeks prior to screening.
* MS/H-10. Prior or concomitant use of cytokine therapy or intravenous immunoglobulins in the 3 months prior to screening.
* MS/H-11. Prior use of alemtuzumab or cladribine.
* MS/H-12. Prior use (within 1 year) of fingolimod (Gilenya®) or natalizumab (Tysabri®).
* MS/H-13. Prior use (within 2 years) of mitoxantrone, or other immunosuppressant agents such as azathioprine, cyclophosphamide, cyclosporine, methotrexate or mycophenolate mofetil.
* MS/H-14. Prior treatment with teriflunomide or leflunomide, unless successful wash-out, confirmed by plasma concentration of < 0.02 μg/ml.
* MS/H-15. Prior use of any investigational drug in the 6 months preceding screening.
* MS/H-16. Pregnant or breast-feeding women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Expression of lymphocyte phenotypic surface markers in dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis. | 0, 8, 16 and 24 weeks after initiation of investigational treatment (week 0)
Expression of lymphocyte phenotypic surface markers in dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis and untreated healthy subjects. | 0, 8, 16 and 24 weeks after initiation of investigational treatment (week 0)

SECONDARY OUTCOMES:
T cell effector functions in terms of cytokine production of CD4+ and CD8+ in dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis. | 0, 8, 16 and 24 weeks after initiation of investigational treatment (week 0)
T cell effector functions in terms of cytokine production of CD4+ and CD8+ in dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis and untreated healthy subjects. | 0, 8, 16 and 24 weeks after initiation of investigational treatment (week 0)
Migratory capacity of immune cells (percentage of migrated cells) in dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis. | 0 and 24 weeks after initiation of investigational treatment (week 0)
Migratory capacity of immune cells (percentage of migrated cells) in dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis and untreated healthy subjects. | 0 and 24 weeks after initiation of investigational treatment (week 0)
Mitochondrial energy metabolism of T cells upon dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis. | 0 and 24 weeks after initiation of investigational treatment (week 0)
Mitochondrial energy metabolism of T cells upon dimethyl fumarate (Tecfidera®)-treated patients with relapsing-remitting multiple sclerosis and untreated healthy subjects. | 0 and 24 weeks after initiation of investigational treatment (week 0)

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Klotz, Prof. Dr., Principal Investigator — University Hospital Muenster
Locations (6):
- Germany (6):
  - Neurologisches Studienzentrum Dr. Schmidt/Dr. Neudecker/ Dr. Viehbahn/Dr. Kronenberger, Bonn
  - Neurologische Gemeinschaftspraxis im Bienenkorbhaus, Frankfurt am Main
  - Neurologische Univ.-Klinik, Heidelberg
  - Klinik und Poliklinik für Neurologie, Universitätsklinikum Mainz, Mainz
  - University Hospital Muenster, Department of Neurology, Münster
  - MVZ-Neurologie Klinikum Osnabrück GmbH, Osnabrück